CLINICAL TRIAL: NCT02750709
Title: A Single Center, Single-Dose, Open-Label, Laboratory-Blind, Randomized, Three-Period Crossover Study to Determine the Bioequivalence of Two Oral Formulations Containing of Nitisinone 10 mg Compared to the Reference Formulation Orfadin 10 mg in at Least 18 Healthy Male and Female Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Two Nitisinone Formulations Compared to Orfadin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cycle Pharmaceuticals Ltd. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CT-001; PXL225418 (Other: PAREXEL (Clinical Trial Unit))
Record Dates: First submitted 2016-04-20; First posted 2016-04-25 (Estimated); Results first posted 2016-12-13 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-02

CONDITIONS: Hereditary Tyrosinemia, Type I
Keywords: HT-1; Tyrosinemia; Nitisinone; Bioequivalence; Healthy Volunteer; Orfadin
MeSH Terms: conditions — Tyrosinemias | interventions — nitisinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment Sequence A (TP 1) - B (TP 2) - C (Reference) (Experimental): Subjects will receive a single 10 mg tablet of Nitisinone 10 mg Tablet (Test Product 1) in treatment period 1, 10 mg tablet of Nitisinone 10 mg Tablet High Compritol (Test Product 2) in treatment period 2, and 10 mg hard capsule of Orfadin (Reference) in treatment period 3 under fasting conditions. Each treatment period will be separated by at least 23 calendar days of washout period.
  Interventions: Drug: Nitisinone; Drug: Nitisinone 10 mg Tablet High Compritol; Drug: Orfadin
- Treatment Sequence A (TP 1) - C (Reference) - B (TP 2) (Experimental): Subjects will receive a single 10 mg tablet of Nitisinone 10 mg Tablet (Test Product 2) in treatment period 1, 10 mg hard capsule of Orfadin (Reference) in treatment period 2, and 10 mg tablet of Nitisinone 10 mg Tablet High Compritol (Test Product 2) in treatment period 3 under fasting conditions. Each treatment period will be separated by at least 23 calendar days of washout period.
  Interventions: Drug: Nitisinone; Drug: Nitisinone 10 mg Tablet High Compritol; Drug: Orfadin
- Treatment Sequence B (TP 2) - A (TP 1) - C (Reference) (Experimental): Subjects will receive a single 10 mg tablet of Nitisinone 10 mg Tablet High Compritol (Test Product 2) in treatment period 1, 10 mg tablet of Nitisinone 10 mg Tablet (Test Product 1) in treatment period 2, and 10 mg hard capsule of Orfadin (Reference) in treatment period 3 under fasting conditions. Each treatment period will be separated by at least 23 calendar days of washout period.
  Interventions: Drug: Nitisinone; Drug: Nitisinone 10 mg Tablet High Compritol; Drug: Orfadin
- Treatment Sequence B (TP 2) - C (Reference) - A (TP 1) (Experimental): Subjects will receive a single 10 mg tablet of Nitisinone 10 mg Tablet High Compritol (Test Product 2) in treatment period 1, 10 mg hard capsule of Orfadin (Reference) in treatment period 2, and 10 mg tablet of Nitisinone 10 mg Tablet (Test Product 1) in treatment period 3, and under fasting conditions. Each treatment period will be separated by at least 23 calendar days of washout period.
  Interventions: Drug: Nitisinone; Drug: Nitisinone 10 mg Tablet High Compritol; Drug: Orfadin
- Treatment Sequence C (Reference) - A (TP 1) - B (TP 2) (Experimental): Subjects will receive a single 10 mg hard capsule of Orfadin (Reference) in treatment period 1, 10 mg tablet of Nitisinone 10 mg Tablet (Test Product 1) in treatment period 2, and 10 mg tablet of Nitisinone 10 mg Tablet High Compritol (Test Product 2) in treatment period 3 under fasting conditions. Each treatment period will be separated by at least 23 calendar days of washout period.
  Interventions: Drug: Nitisinone; Drug: Nitisinone 10 mg Tablet High Compritol; Drug: Orfadin
- Treatment Sequence C (Reference) - B (TP 2) - A (TP 1) (Experimental): Subjects will receive a single 10 mg hard capsule of Orfadin (Reference) in treatment period 1, 10 mg tablet of Nitisinone 10 mg Tablet High Compritol (Test Product 2) in treatment period 2, 10 mg tablet of Nitisinone 10 mg Tablet (Test Product 1) in treatment period 3 under fasting conditions. Each treatment period will be separated by at least 23 calendar days of washout period.
  Interventions: Drug: Nitisinone; Drug: Nitisinone 10 mg Tablet High Compritol; Drug: Orfadin

INTERVENTIONS:
Drug: Nitisinone — A single oral dose of Nitisinone 10 mg tablet will be administered in fasted state.
Drug: Nitisinone 10 mg Tablet High Compritol — A single oral dose of Nitisinone 10 mg High Compritol tablet will be administered in fasted state.
Drug: Orfadin — A single oral dose of Orfadin 10 mg hard capsule will be administered in fasted state.

SUMMARY:
The purpose of this study is to determine whether Nitisinone 10 mg Tablets (Test Product 1 (TP1)) and Nitisinone 10 mg Tablets High Compritol (Test Product 2 (TP2)) are bioequivalent to the reference product Orfadin 10 mg capsules.

DETAILED DESCRIPTION:
The specific aim is to conduct a randomized, single dose, three-period cross-over bioequivalence (BE) study in at least 18 healthy male and female subjects at a single study center to evaluate the in vivo performance of Nitisinone 10 mg Tablet (Test Product 1) and Nitisinone 10 mg Tablet High Compritol (Test Product 2) to the reference product Orfadin 10 mg capsules.

The pharmacokinetics (PK) of Test Product 1 and 2 compared to the reference product, will be determined and compared in healthy volunteers.

The modified version of Nitisinone Tablet (Test Product 2, higher glyceryl dibehenate (Compritol 888)) was administered to determine the acceptance limit of the dissolution profile for Nitisinone tablets with a longer dissolution time (Test Product 2) since the dissolution time of Nitisinone tablets (Test Product 1) lengthened over time under accelerated study conditions. The hypothesis is that should bioequivalence between Test Product 1 and Test Product 2 be demonstrated then it is concluded that the prolonged dissolution time had no impact on the bioequivalence of Nitisinone tablets.

A total of 24 healthy female and male volunteers (age 18 to 55 years old) will be entered into the study. Volunteers will be determined to be free of significant medical conditions as assessed by medical history, physical examination, and blood and urine tests. Volunteers will be randomly allocated to receive one of the three treatment sequence groups and, on each occasion, receive one of the following: Nitisinone 10 mg Tablet, Nitisinone 10 mg High Compritol Tablet and Orfadin 10 mg hard capsules (reference listed drug, (RLD)). There will be a minimum 23 calendar days washout between treatments. Blood samples will be collected at pre-dose (0 hours) and at 15 minutes, 30 minutes, 1 hour, 2 hours, 2 hours and 30 minutes, 3 hours, 3 hours and 30 minutes, 4 hours, 5 hours, 6 hours, 7 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 96 hours and 120 hours post-dose (total: 21 samples per treatment period).

The primary endpoints will be the maximum blood concentration (Cmax) and the area under the curve (AUC) from time zero to 120 hours post-dose.

For the FDA, bioequivalence of the test and reference products will be assessed on the basis of the 90% confidence intervals for estimates of the geometric mean ratios between the primary PK parameters of the test and reference products using an analysis of variance considering the bioequivalence range of 80.00% to 125.00% for Cmax and AUC(0-120).

For Health Canada, bioequivalence of the test and reference products will be assessed on the basis of the 90% confidence interval for estimate of the geometric mean ratio between the primary PK parameter AUC(0-120) of the test and reference products using an analysis of variance considering the bioequivalence range of 80.00% to 125.00% and the point estimate of the geometric mean ratio of the primary PK parameter Cmax considering the bioequivalence range of 80.00% to 125.00%.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18.5 and 30 kg/m2 (inclusive).
* Body mass not less than 50 kg.
* Medical history, vital signs, physical examination, standard 12-lead electrocardiogram (ECG) and laboratory investigations must be clinically acceptable or within laboratory reference ranges for the relevant laboratory tests, unless the investigator considers the deviation to be irrelevant for the purpose of the study.
* Non-smokers.
* Females, if:

Not of childbearing potential, e.g., has been surgically sterilized, undergone a hysterectomy, amenorrhea for ≥ 12 months and considered post-menopausal,

Note: In postmenopausal women, the value of the serum pregnancy test may be slightly increased. This test will be repeated to confirm the results. If there is no increase indicative of pregnancy, the female will be included in the study.

OR

Of childbearing potential, the following conditions are to be met:

* Negative pregnancy test
* If this test is positive, the subject will be excluded from the study. In the rare circumstance that a pregnancy is discovered after the subject received Investigational Medicinal Product (IMP), every attempt must be made to follow her to term.
* Not lactating
* Abstaining from sexual activity (if this is the usual lifestyle of the subject) or must agree to use an accepted method of contraception, and agree to continue with the same method throughout the study

Examples of reliable methods of contraception include non-hormonal intrauterine device, and barrier methods combined with an additional contraceptive method.

In this study the concomitant use of hormonal contraceptives is NOT allowed.

Other methods, if considered by the investigator as reliable, will be accepted.

* Written consent given for participation in the study.

Exclusion Criteria:

* Evidence of psychiatric disorder, antagonistic personality, poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
* Current alcohol use > 21 units of alcohol per week for males and > 14 units of alcohol per week for females.
* Consumption of more than 5 cups of coffee (or equivalent amounts of caffeine) per day.
* Regular exposure to substances of abuse (other than alcohol) within the past year.
* Use of any medication, prescribed or over-the-counter or herbal remedies, within 2 weeks before the first administration of IMP except if this will not affect the outcome of the study in the opinion of the investigator. In this study the concomitant use of hormonal contraceptives is NOT allowed.
* Participation in another study with an experimental drug, where the last administration of the previous IMP was within 8 weeks (or within 10 elimination half-lives for chemical entities or 2 elimination half-lives for antibodies or insulin), whichever is the longer) before administration of IMP in this study, at the discretion of the investigator.
* Treatment within the previous 3 months before the first administration of IMP with any drug with a well-defined potential for adversely affecting a major organ or system.
* A major illness during the 3 months before commencement of the screening period.
* History of hypersensitivity or allergy to the IMP or its excipients or any related medication.
* History of bronchial asthma or any other bronchospastic disease.
* History of convulsions.
* History of porphyria.
* Relevant history or laboratory or clinical findings indicative of acute or chronic disease, likely to influence study outcome.
* Donation or loss of blood equal to or exceeding 500 mL during the 8 weeks before the first administration of IMP.
* Diagnosis of hypotension made during the screening period.
* Diagnosis of hypertension made during the screening period or current diagnosis of hypertension.
* Resting pulse of > 100 beats per minute or < 40 beats per minute during the screening period, either supine or standing.
* Positive testing for human immunodeficiency virus (HIV), Hepatitis B and Hepatitis C.
* Positive urine screen for drugs of abuse. In case of a positive result the urine screen for drugs of abuse may be repeated once at the discretion of the investigator.
* Positive urine screen for tobacco use.
* Positive pregnancy test.
* Female subjects that are pregnant or breastfeeding.
* Difficulty in swallowing.
* Any specific investigational product safety concern.
* Vulnerable subjects, e.g. persons in detention.
* Subjects with current keratopathy, or other clinically significant abnormalities found by slit-lamp examination (cataracts) at the discretion of the investigator.
* Concomitant use of medications that are metabolized by CYP2C9 (ibuprofen, diclofenac and indomethacin).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: André Nell, Principal Investigator — Bloemfontein Early Phase Clinical Unit, PAREXEL Internation (South Africa)
Locations (1):
- Bloemfontein Early Phase Clinical Unit, PAREXEL International (South Africa), Bloemfontein, Free State, South Africa

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1
Arm/Group | Treatment Sequence A (TP 1) - B (TP 2) - C (Reference) | Treatment Sequence A (TP 1) - C (Reference) - B (TP 2) | Treatment Sequence B (TP 2) - A (TP 1) - C (Reference) | Treatment Sequence B (TP 2) - C (Reference) - A (TP 1) | Treatment Sequence C (Reference) - A (TP 1) - B (TP 2) | Treatment Sequence C (Reference) - B (TP 2) - A (TP 1)
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Period: Treatment Period 2
Arm/Group | Treatment Sequence A (TP 1) - B (TP 2) - C (Reference) | Treatment Sequence A (TP 1) - C (Reference) - B (TP 2) | Treatment Sequence B (TP 2) - A (TP 1) - C (Reference) | Treatment Sequence B (TP 2) - C (Reference) - A (TP 1) | Treatment Sequence C (Reference) - A (TP 1) - B (TP 2) | Treatment Sequence C (Reference) - B (TP 2) - A (TP 1)
Started | 4 | 4 | 4 | 4 | 4 | 3
Completed | 4 | 4 | 4 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Treatment Sequence A (TP 1) - B (TP 2) - C (Reference) | Treatment Sequence A (TP 1) - C (Reference) - B (TP 2) | Treatment Sequence B (TP 2) - A (TP 1) - C (Reference) | Treatment Sequence B (TP 2) - C (Reference) - A (TP 1) | Treatment Sequence C (Reference) - A (TP 1) - B (TP 2) | Treatment Sequence C (Reference) - B (TP 2) - A (TP 1)
Started | 4 | 4 | 4 | 4 | 4 | 3
Completed | 4 | 4 | 4 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 19
Race/Ethnicity, Customized [Number; unit: Participants]
  Black | 15
  Caucasian | 7
  Coloured | 1
  Mixed Race | 1
Region of Enrollment [Number; unit: participants]
  South Africa | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0, 0.25, 0.50, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96 and 120 hours
Population: All subjects for whom the primary PK parameters Cmax and AUC(0-120) could be calculated for at least 2 treatment periods (where one of the treatment periods is the Reference product), and who had no major protocol deviations thought to impact on the analysis of the PK data were included in the statistical PK analysis for the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Treatment Period 1: Nitisinone Tablet, 10 mg
- Treatment Period 2: Nitisinone Tablet (High Compritol), 10 mg
- Reference Product: ORFADIN® hard capsule, 10 mg
Arm/Group | Treatment Period 1 | Treatment Period 2 | Reference Product
Number analyzed (Participants) | 23 | 23 | 23
ng/mL | 1137.40 (17.9) | 1080.69 (24.2) | 1168.71 (22.6)

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve, From Time Zero to 120 Hours Post-dose (AUC(0-120))
Time Frame: 0, 0.25, 0.50, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96 and 120 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Treatment Period 1 | Treatment Period 2 | Reference Product
Number analyzed (Participants) | 23 | 23 | 23
hr*ng/mL | 66220.91 (19.0) | 61883.52 (23.1) | 66199.76 (18.7)

3. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve, From Time Zero to 72 Hours Post-dose (AUC(0-72))
Time Frame: 0, 0.25, 0.50, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Treatment Period 1 | Treatment Period 2 | Reference Product
Number analyzed (Participants) | 23 | 23 | 23
hr*ng/mL | 49448.49 (19.8) | 46401.12 (37.6) | 49582.69 (19.2)

4. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve, With Extrapolation to Infinity (AUC(0-∞)
Time Frame: 0, 0.25, 0.50, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96 and 120 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Treatment Period 1 | Treatment Period 2 | Reference Product
Number analyzed (Participants) | 23 | 23 | 23
hr*ng/mL | 91226.27 (26.6) | 83245.33 (37.0) | 89394.35 (23.7)

5. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax)
Time Frame: 0, 0.25, 0.50, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96 and 120 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | Treatment Period 1 | Treatment Period 2 | Reference Product
Number analyzed (Participants) | 23 | 23 | 23
hr | 3.00 [2.00 to 5.00] | 3.00 [1.00 to 7.00] | 2.50 [0.50 to 8.00]

6. Secondary Outcome: Terminal Elimination Rate Constant (λz)
Time Frame: 0, 0.25, 0.50, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96 and 120 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hr
Arm/Group | Treatment Period 1 | Treatment Period 2 | Reference Product
Number analyzed (Participants) | 23 | 23 | 23
1/hr | 0.011 (29.1) | 0.012 (20.6) | 0.012 (25.2)

7. Secondary Outcome: Apparent Terminal Half-life (t1/2)
Time Frame: 0, 0.25, 0.50, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72, 96 and 120 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Treatment Period 1 | Treatment Period 2 | Reference Product
Number analyzed (Participants) | 23 | 23 | 23
hr | 61.42 (29.1) | 58.41 (20.6) | 59.43 (25.2)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the period of the study (December 2015 - January 2016).
Description: 24 subjects were entered in to the study and randomly assigned to treatment sequence according to randomization schedule before first administration of the Investigational Medicinal Product (IMP). One subject was withdrawn from the study after Treatment Period 1 (Reference Product) because they vomited within 2 times median Tmax. As a result, 24 subjects completed dosing of Reference Product and 23 subjects completed the study.
Groups:
- Test Product 1: Nitisinone Tablet, 10 mg
- Test Product 2: Nitisinone Tablet (High Compritol), 10 mg
Arm/Group | Test Product 1 | Test Product 2 | Reference Product
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 1/23 | 1/23 | 2/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product 1 (N=23) | Test Product 2 (N=23) | Reference Product (N=24)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Itching Fingers (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Vaso Vagal Attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No